CLINICAL TRIAL: NCT02884245
Title: Interest of Estrogen Scheduling Before Ovarian Stimulation With Corifollitropin Alfa in Women Older Than 38 Years Old Undergoing in Vitro Fertilization
Brief Title: Interest of Estrogen Scheduling Before Ovarian Stimulation With Corifollitropin Alfa
Acronym: PRESCORI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Anne GUIVARC'H-LEVEQUE, Reproductive Endocrinologist, Centre Hospitalier Intercommunal Creteil
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRESCORI
Record Dates: First submitted 2016-08-22; First posted 2016-08-30 (Estimated); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Infertility
Keywords: Fertility; Reproductive processes; In vitro fertilization; Intracytoplasmic sperm injection; Estrogens; Follicule Stimulating Hormon
MeSH Terms: conditions — Infertility | interventions — Estrogens

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm E2: With estrogens pretreatment (Experimental): The estrogens pretreatment will began between the day 20 and the day 24 of an ovarian cycle and should be continued until Wednesday beyond the onset of menses
  Interventions: Drug: Estrogens
- Arm S: without estrogens pretreatment (No Intervention): No estrogen pretreatment will be delivered

INTERVENTIONS:
Drug: Estrogens — The estrogens pretreatment will began between the day 20 and the day 24 of an ovarian cycle and should be continued until Wednesday beyond the onset of menses
  Arms: Arm E2: With estrogens pretreatment

SUMMARY:
E2 given in late luteal phase can be extended beyond the onset of menses for a period of at least eight days before the start of the stimulation, allowing scheduling of stimulation in order to limit oocytes retrievals during weekends .

Administration of corifollitropin alfa, a Follicule stimulating Hormone (FSH) with extended release kinetics, seems particularly interesting for a synchronous recruitment of follicles after homogenization of the cohort.

The objective of this study is to evaluate the impact on the response to ovarian stimulation with corifollitropin alfa of E2 scheduling versus no scheduling for women over 38 years, age at which declining of ovarian reserve usually begins. The management of these patients in terms of organization of the center is also evaluated.

The scheduling of IVF cycles represents a double benefit. On one hand, to enable a "synchronization" of the follicular cohort for a best response and a higher number of mature oocytes. On the other hand, a more efficient organization for both the center (avoiding retrievals on weekends and public holidays, organize and distribute equally the activity, reduce cost operations) and couples (personal and professional organization).

DETAILED DESCRIPTION:
With advanced age, ovarian reserve decreases, follicular cohort becomes heterogeneous under the influence of higher FSH rise in late luteal phase. It has been shown that estrogens (E2) taken in the late luteal phase homogenized follicular cohort by inhibiting inter cycle FSH peak ,and that this inhibition is immediately reversible after discontinuation of treatment .

E2 given in late luteal phase can also be extended beyond the onset of menses for a period of at least eight days before the start of the stimulation, allowing scheduling of stimulation in order to limit oocytes retrievals during weekends . A prospective randomized study comparing E2 scheduling and no scheduling has shown that there was no difference in birth rate in a population of normo-responders women . While in these patients, the number of oocytes was not different in the two arms, a recent pilot study founded a significant increase in the number of oocytes retrieved after E2 luteal phase priming compared to the absence of priming in a population of poor responders .

In 2013, a report of the French governmental BioMedicine Agency warned about the thrombo-embolic risk associated with the use of the contraceptive pill for IVF scheduling, especially in women over 35.

Administration of corifollitropin alfa, an FSH with extended release kinetics, seems particularly interesting for a synchronous recruitment of follicles after homogenization of the cohort. In the Pursue study, an equivalent efficacy has been shown with the daily administration of 300 IU FSH and corifollitropin alfa in patients over 35 years .

The objective of this study is to evaluate the impact of the response to ovarian stimulation with corifollitropin alfa of E2 scheduling versus no scheduling for women over 38 years, age at which declining of ovarian reserve usually begins. The management of these patients in terms of organization of the center is also evaluated.

The scheduling of IVF cycles represents a double benefit. On one hand, to enable a "synchronization" of the follicular cohort for a best response and a higher number of mature oocytes. On the other hand, a more efficient organization for both the center (avoiding retrievals on weekends and public holidays, organize and distribute equally the activity, reduce cost operations) and couples (personal and professional organization). This can be done with pills but there are controversial data on its impact on the chances of birth. It has been shown that estrogen scheduling provides opportunities for success equivalent to the absence of scheduling for patients with good prognosis . If this study confirms the initial hypothesis, it will show that a less favorable public can profit from the benefits of scheduling by estrogen on both the organization of the attempt and the chances of pregnancy through better ovarian response.

ELIGIBILITY:
Inclusion Criteria:

* Patient of 38 years or more
* Planned in invitro fertilization or intracytoplasmic sperm injection rank 1 or 2 (rank = retrieval with transfer)
* With regular cycles from 26 to 35 days
* Weight > 50 kg and body mass index< or equal to 32
* Affiliation to the general system of French social security and reimbursement for fertility problems

Exclusion Criteria:

* Irregular cycles and/or polycystic ovarian syndrome
* Previous History of ovarian hyperstimulation syndrome
* Rank puncture > 2
* Uterine malformation
* Presence of hydrosalpinges
* Endometriosis stage III or IV

Ages: 38 Years to 47 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 334 (Actual)
Dates: Start 2016-11-04 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2023-01-04 (Actual)

PRIMARY OUTCOMES:
Number of selected oocytes | At time of ovarian puncture

SECONDARY OUTCOMES:
Number of days of pretreatment | From inclusion visit date to the beginning of stimulation, up to 15 days
Cancellation rate | From date of inclusion visit until the date of embryo transfer, up to 90 days
Number of days of antagonist | From date of stimulation until the date of the trigger, up to 30 days
The day of the trigger | At time of the trigger
Estradiol rate | 8 days from the beginning of stimulation and the day of the trigger
Luteinizing hormone rate | 8 days from the beginning of stimulation and the day of the trigger
Progesterone rate | 8 days from the beginning of stimulation and the day of the trigger
Follicles number > 10 mm | 8 days from the beginning of stimulation
Follicles number > 14 mm | From 1 day before the day of trigger or the day of trigger
Number of oocytes in metaphase 2 | At time of ovarian puncture
Total number of embryos with good quality | At time of fertilization procedure
early pregnancy | 14 days after embryo transfer
  Beta Human chorionic gonadotropin>100 U/l
ongoing pregnancy rate | 12 weeks after embryo transfer
  on ultrasound procedure
miscarriage before 12 weeks of amenorrhea | From embryo transfer to 12 weeks after embryo transfer

CONTACTS AND LOCATIONS:
Overall Officials: Anne GUIVARC'H - LEVEQUE, MD, Principal Investigator — Clinique de la Sagesse; Isabelle CEDRIN - DURNERIN, MD, Principal Investigator — CHU Jean Verdier - APHP; Nathalie MASSIN, MD, Principal Investigator — CHI Créteil
Locations (3):
- France (3):
  - Hôpital Jean Verdier, Bondy
  - CHI Creteil, Créteil
  - Clinique de la Sagesse, Rennes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Blockeel C, Engels S, De Vos M, Haentjens P, Polyzos NP, Stoop D, Camus M, Devroey P. Oestradiol valerate pretreatment in GnRH-antagonist cycles: a randomized controlled trial. Reprod Biomed Online. 2012 Mar;24(3):272-80. doi: 10.1016/j.rbmo.2011.11.012. Epub 2011 Nov 30. PMID 22296973
- [Background] Boostanfar R, Shapiro B, Levy M, Rosenwaks Z, Witjes H, Stegmann BJ, Elbers J, Gordon K, Mannaerts B; Pursue investigators. Large, comparative, randomized double-blind trial confirming noninferiority of pregnancy rates for corifollitropin alfa compared with recombinant follicle-stimulating hormone in a gonadotropin-releasing hormone antagonist controlled ovarian stimulation protocol in older patients undergoing in vitro fertilization. Fertil Steril. 2015 Jul;104(1):94-103.e1. doi: 10.1016/j.fertnstert.2015.04.018. Epub 2015 May 21. PMID 26003273
- [Background] Cedrin-Durnerin I, Bstandig B, Parneix I, Bied-Damon V, Avril C, Decanter C, Hugues JN. Effects of oral contraceptive, synthetic progestogen or natural estrogen pre-treatments on the hormonal profile and the antral follicle cohort before GnRH antagonist protocol. Hum Reprod. 2007 Jan;22(1):109-16. doi: 10.1093/humrep/del340. Epub 2006 Aug 26. PMID 16936304
- [Background] Cedrin-Durnerin I, Guivarc'h-Leveque A, Hugues JN; Groupe d'Etude en Medecine et Endocrinologie de la Reproduction. Pretreatment with estrogen does not affect IVF-ICSI cycle outcome compared with no pretreatment in GnRH antagonist protocol: a prospective randomized trial. Fertil Steril. 2012 Jun;97(6):1359-64.e1. doi: 10.1016/j.fertnstert.2012.02.028. Epub 2012 Mar 28. PMID 22464760
- [Background] Chang X, Wu J. Effects of luteal estradiol pre-treatment on the outcome of IVF in poor ovarian responders. Gynecol Endocrinol. 2013 Mar;29(3):196-200. doi: 10.3109/09513590.2012.736558. Epub 2012 Nov 30. PMID 23194136
- [Background] Escriva AM, Diaz-Garcia C, Monterde M, Rubio JM, Pellicer A. Antral Follicle Priming Before Intracytoplasmic Sperm Injection in Previously Diagnosed Low Responders: A Randomized Controlled Trial (FOLLPRIM). J Clin Endocrinol Metab. 2015 Jul;100(7):2597-605. doi: 10.1210/jc.2015-1194. Epub 2015 May 8. PMID 25955224
- [Background] Fanchin R, Salomon L, Castelo-Branco A, Olivennes F, Frydman N, Frydman R. Luteal estradiol pre-treatment coordinates follicular growth during controlled ovarian hyperstimulation with GnRH antagonists. Hum Reprod. 2003 Dec;18(12):2698-703. doi: 10.1093/humrep/deg516. PMID 14645194
- [Background] Guivarc'h-Leveque A, Homer L, Arvis P, Broux PL, Moy L, Priou G, Vialard J, Colleu D, Dewailly D. Programming in vitro fertilization retrievals during working days after a gonadotropin-releasing hormone antagonist protocol with estrogen pretreatment: does the length of exposure to estradiol impact on controlled ovarian hyperstimulation outcomes? Fertil Steril. 2011 Oct;96(4):872-6. doi: 10.1016/j.fertnstert.2011.07.1138. Epub 2011 Aug 24. PMID 21868004
- [Background] Hauzman EE, Zapata A, Bermejo A, Iglesias C, Pellicer A, Garcia-Velasco JA. Cycle scheduling for in vitro fertilization with oral contraceptive pills versus oral estradiol valerate: a randomized, controlled trial. Reprod Biol Endocrinol. 2013 Sep 28;11:96. doi: 10.1186/1477-7827-11-96. PMID 24074027
- [Background] Nielsen AP, Korsholm AS, Lemmen JG, Sylvest R, Sopa N, Nyboe Andersen A. Selective use of corifollitropin for controlled ovarian stimulation for IVF in patients with low anti-Mullerian hormone. Gynecol Endocrinol. 2016 Aug;32(8):625-628. doi: 10.3109/09513590.2016.1147548. Epub 2016 Feb 18. PMID 26891977
- [Background] Polyzos NP, De Vos M, Corona R, Vloeberghs V, Ortega-Hrepich C, Stoop D, Tournaye H. Addition of highly purified HMG after corifollitropin alfa in antagonist-treated poor ovarian responders: a pilot study. Hum Reprod. 2013 May;28(5):1254-60. doi: 10.1093/humrep/det045. Epub 2013 Feb 26. PMID 23442756
- [Background] Reynolds KA, Omurtag KR, Jimenez PT, Rhee JS, Tuuli MG, Jungheim ES. Cycle cancellation and pregnancy after luteal estradiol priming in women defined as poor responders: a systematic review and meta-analysis. Hum Reprod. 2013 Nov;28(11):2981-9. doi: 10.1093/humrep/det306. Epub 2013 Jul 25. PMID 23887073
- [Derived] Cedrin-Durnerin I, Carton I, Massin N, Chevalier N, Dubourdieu S, Bstandig B, Michelson X, Goro S, Jung C, Guivarc'h-Leveque A. Pretreatment with luteal estradiol for programming antagonist cycles compared to no pretreatment in advanced age women stimulated with corifollitropin alfa: a non-inferiority randomized controlled trial. Hum Reprod. 2024 Sep 1;39(9):1979-1986. doi: 10.1093/humrep/deae167. PMID 39008826